CLINICAL TRIAL: NCT06904014
Title: Exploratory Study on the Efficacy and Safety of Sintilimab Combined With Lenvatinib and HAIC for Neoadjuvant Therapy of Borderline Resectable Hepatocellular Carcinoma
Brief Title: Efficacy and Safety of Sintilimab Combined With Lenvatinib and HAIC for Neoadjuvant Therapy of Borderline Resectable HCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei ZHAO (Other)
Responsible Party: Sponsor-Investigator, Lei ZHAO, Doctor, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2023-110-01
Record Dates: First submitted 2025-03-21; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HCC
MeSH Terms: interventions — sintilimab; lenvatinib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental：Sintilimab+ Lenvatinib+HAIC+surgery (Experimental): the experimental group received 200 mg of sintilimab by intravenous infusion on the first day of every 3 weeks. Lenvatinib 8 mg was orally administered once daily, combined with the HAIC-FOLFOX regimen. After two cycles, the patients' conditions were evaluated for surgery
  Interventions: Procedure: HAIC; Drug: Sintilimab; Drug: Lenvatinib; Procedure: surgery
- Control (Other): surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: HAIC — FOLFOX-hepatic artery infusion
  Arms: Experimental：Sintilimab+ Lenvatinib+HAIC+surgery
Drug: Sintilimab — 200mg, ivgtt, D1, Q3W
  Arms: Experimental：Sintilimab+ Lenvatinib+HAIC+surgery
Drug: Lenvatinib — 8 mg，qd，D1-D21,Q3W
  Arms: Experimental：Sintilimab+ Lenvatinib+HAIC+surgery
Procedure: surgery — surgery

SUMMARY:
This study is a single-center, randomized controlled exploratory Phase II clinical trial, aiming to assess the efficacy and safety of sintilimab combined with lenvatinib and HAIC for two cycles followed by surgery compared with direct surgery in patients with borderline resectable hepatocellular carcinoma.

After signing the informed consent and meeting the inclusion and exclusion criteria, the eligible subjects were randomly divided into the experimental group and the control group:

* Subjects in the experimental group received 200 mg of sintilimab by intravenous infusion on the first day of every 3 weeks. Lenvatinib 8 mg was orally administered once daily, combined with the HAIC-FOLFOX regimen. After two cycles, the patients' conditions were evaluated for surgery.
* Subjects in the control group underwent surgery directly.

Both groups of subjects received sintilimab monotherapy as adjuvant treatment for half a year (a total of 8 cycles) after surgery. The treatment was terminated if there was disease recurrence, death, intolerable toxicity, withdrawal of informed consent, initiation of new anti-tumor treatment, or other reasons stipulated in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent before the implementation of any trial-related procedures.
2. Male or female, aged ≥18 years and ≤70 years.
3. ECOG PS score of 0-2.
4. Diagnosed with HCC according to the Diagnosis and Treatment Guidelines for Primary Liver Cancer in China (2019 Edition).
5. CNLC stage IIIa, with vascular invasion but no extrahepatic metastasis.
6. Child-Pugh score of A/B.
7. Portal vein tumor thrombus is classified as type 1-2 according to the Japanese VP classification or type I-II according to the Program classification.
8. No previous systemic anti-tumor treatment for hepatocellular carcinoma and eligible for R0 resection.
9. Expected survival time > 3 months.
10. At least one measurable lesion according to RECIST 1.1 or mRECIST criteria.
11. Adequate organ and bone marrow function, as follows:

1) Blood routine: absolute neutrophil count (ANC) ≥ 1.5×109/L; platelet count (PLT) ≥ 75×109/L; hemoglobin content (HGB) ≥ 9.0 g/dL.

2) Liver function: serum total bilirubin (TBIL) ≤ 3×ULN; alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 5×ULN; serum albumin ≥ 28 g/L.

3) Renal function: serum creatinine (Cr) ≤ 1.5×ULN or clearance of creatinine (CCr) ≥ 50 mL/min (Cockcroft-Gault formula); urine routine test shows urine protein < 2+; for patients with urine protein ≥ 2+ at baseline, 24-hour urine collection is required and 24-hour urine protein quantification < 1 g.

4) Coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5×ULN.

12. For patients with acute or chronic active hepatitis B or C, continuous antiviral treatment is required during the study period.

13. For female subjects of childbearing age, a urine or serum pregnancy test must be negative within 3 days before the first administration of the study drug (day 1 of cycle 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Non-childbearing age females are defined as those who have been postmenopausal for at least 1 year, or have undergone surgical sterilization or hysterectomy.

14. If there is a risk of pregnancy, all subjects (regardless of gender) must use a contraceptive method with a failure rate of less than 1% throughout the treatment period until 120 days after the last administration of the study drug (or 180 days after the last administration of chemotherapy drugs). Expected survival time ≥ 12 weeks.

Exclusion Criteria:

1. Previously histologically/cytologically confirmed liver cancer with components such as fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, etc.
2. History of hepatic encephalopathy or liver transplantation.
3. Clinical symptoms requiring drainage of pleural effusion, ascites, or pericardial effusion.
4. Acute or chronic active hepatitis B or C infection, with HBV DNA > 2000 IU/ml or 104 copies/ml; HCV RNA > 103 copies/ml; positive for both hepatitis B surface antigen (HbsAg) and anti-HCV antibody.
5. Central nervous system metastasis.
6. Esophageal or gastric variceal bleeding events due to portal hypertension within the past 6 months. Known severe (G3) varices on endoscopy within 3 months before the first dose. Evidence of portal hypertension (including splenomegaly on imaging), and high bleeding risk as assessed by the investigator.
7. Any life-threatening bleeding events within the past 3 months, including those requiring blood transfusion, surgery or local treatment, or continuous drug treatment.
8. Venous or arterial thromboembolic events within the past 6 months, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis or any other serious thromboembolic events. Patients with stable thrombosis after conventional anticoagulation treatment, such as those with implanted venous access ports or catheter-related thrombosis, or superficial vein thrombosis, are excluded. Prophylactic use of low-dose low-molecular-weight heparin (e.g., enoxaparin 40 mg/day) is allowed.
9. Use of aspirin (> 325 mg/day) or other known platelet function inhibitors such as dipyridamole or clopidogrel for 10 consecutive days within 2 weeks before the first dose.
10. Uncontrolled hypertension, with systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg after optimal medical treatment, or history of hypertensive crisis or hypertensive encephalopathy.
11. Symptomatic congestive heart failure (NYHA class II-IV). Symptomatic or poorly controlled arrhythmia. History of congenital long QT syndrome or corrected QTc > 500 ms (calculated using the Fridericia method) at screening.
12. Severe bleeding tendency or coagulation disorders, or currently undergoing thrombolytic therapy.
13. History of gastrointestinal perforation and/or fistula within the past 6 months, history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive intestinal resection (partial colectomy or extensive small bowel resection, concurrent with chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea.
14. Received radiotherapy within 3 weeks before the first dose. For patients who received radiotherapy more than 3 weeks before the first dose, all of the following conditions must be met to be eligible for inclusion: no current radiotherapy-related toxicities, no need for glucocorticoids, and exclusion of radiation pneumonitis, radiation hepatitis, radiation enteritis, etc.
15. History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, or severe lung function impairment.
16. Human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive), or known syphilis infection.
17. Active or poorly controlled severe infection. Severe infection within 4 weeks before the first dose, including but not limited to hospitalization due to infection, bacteremia, or complications of severe pneumonia.
18. Active or poorly controlled autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years before the first dose. Use of replacement therapy (e.g., thyroid hormone, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is allowed. A known history of primary immunodeficiency. Patients with only positive autoimmune antibodies need to be confirmed by the investigator as having no autoimmune disease.
19. Use of immunosuppressive drugs within 4 weeks before the first dose, excluding nasal sprays, inhalation or other local glucocorticoids or physiological doses of systemic glucocorticoids (i.e., no more than 10mg/day of prednisone or equivalent doses of other glucocorticoids), and temporary use of glucocorticoids for the treatment of breathing difficulties due to asthma, chronic obstructive pulmonary disease, etc. is allowed.
20. Receipt of live attenuated vaccines within 4 weeks before the first dose or planned during the study period.
21. Receipt of local treatment for liver cancer within 4 weeks before the first dose.
22. Receipt of traditional Chinese medicine with anti-tumor indications or drugs with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural or ascitic fluid) within 2 weeks before the first dose.
23. Uncontrolled or uncorrectable metabolic disorders or other non-malignant organ diseases or systemic diseases or secondary reactions of cancer that may lead to higher medical risks and/or uncertainty in survival evaluation.
24. Diagnosis of other malignancies within 5 years before the first dose, excluding skin basal cell carcinoma, skin squamous cell carcinoma, and/or in situ carcinoma that have been completely resected. If other malignancies or liver cancer were diagnosed more than 5 years before the first dose, pathological or cytological diagnosis of recurrent or metastatic lesions is required.
25. Previous receipt of any anti-PD-1 antibody, anti-PD-L1/L2 antibody, anti-CTLA4 antibody, or other immunotherapy.
26. Known allergy to any component of sintilimab, lenvatinib, or chemotherapy drugs; or previous severe allergic reactions to other monoclonal antibodies or tyrosine kinase inhibitors.
27. Receipt of treatment in other clinical trials within 4 weeks before the first dose.
28. Pregnant or lactating female patients.
29. Other acute or chronic diseases, mental disorders, or abnormal laboratory test values that may lead to the following results: increased risks associated with study participation or administration of the study drug, or interference with the interpretation of study results, and the patient is judged by the investigator as not eligible to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
One-year disease-free survival rate | From enrollment to the end of treatment at one year
  The 1-year disease-free survival rate (1-year DFS rate) of the experimental group and the control group

SECONDARY OUTCOMES:
disease-free survival（DFS） | From enrollment to the end of treatment，assessed up to 3 years
  The time from enrollment to the first radiological disease recurrence or death (whichever occurred first)
Overall survival (OS) | Up to three years
  as the time from enrollment to the death of the subject for any reason
Pathologic complete response (pCR) | Up to one year
  The proportion of subjects whose postoperative pathological examination did not detect residual cancer cells

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No